CLINICAL TRIAL: NCT05115448
Title: Effect of Bevel Position of the Artery Needle on Puncture Pain and Post-puncture Bleeding Time in Hemodialysis Patients
Brief Title: Effect of Bevel Position of the Artery Needle on Puncture Pain and Post-puncture Bleeding Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07/16/2019
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Pain; Bleeding Time; Arteriovenous Fistula
MeSH Terms: conditions — Pain; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevel Up (Other): In the patients who participated in the study, cannulation was applied to the fistula with the needle direction antegrade and the needle pointing upwards for the first 6 sessions, and the needle direction antegrade and the needle tip facing down for the next 6 sessions. The cannulation procedure was performed by the same nurse for each patient who participated in the study.
  Interventions: Other: Bevel Position
- Bevel Down (Other): In the patients who participated in the study, cannulation was applied to the fistula with the needle direction antegrade and the needle pointing downwards for the next 6 sessions. The cannulation procedure was performed by the same nurse for each patient who participated in the study.
  Interventions: Other: Bevel Position

INTERVENTIONS:
Other: Bevel Position — During 6 dialysis sessions, cannulation was applied to the patients with the direction of the arterial needle in the antegrade direction and the conical tip facing upwards. In the next 6 dialysis sessions, cannulation was applied to the patients in an antegrade direction and with the conical tip facing down.

SUMMARY:
A patient with an arteriovenous fistula (AVF) receiving chronic hemodialysis (HD) treatment is cannulated 312 times a year on average. The patients cannot comply with dialysis treatment and the quality of life is decreased by pain when the fistula cannot be accessed with a single attempt. Sharp pain depends on the tear in the skin, the tissue where the sensitive nerve ends receptive to pain are located, and it is particularly important during AVF puncture. Also, punctures are accompanied by haemorrhages and frequent loss of blood.

DETAILED DESCRIPTION:
The repeated puncture of the AVF leads to a considerable degree of pain, due to the calibre and length of the bevel of fistula needles. When the fistula needle is removed, the small punctures that occur in the entrance area are closed with a thrombus. As a result, scar tissue forms in the entrance area and the surrounding skin, which can lead to the development of stenosis and aneurysm. For this reason, the needle conical tip direction is important in terms of delaying the loss of tissue elasticity and prolonging the use of the intervention area. There are very few studies investigating the effect of the conical tip being up or down on the pain that develops during cannulation in the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* On maintenance hemodialysis three times per week for four hours per session
* Receiving hemodialysis therapy for a least six moths at the time of the study
* Pain level of one or more measured by the Visual Analogue Scale during cannulation
* Able to communicate in Turkish
* Willing to participate to the study

Exclusion Criteria:

* Known to be difficult to enter the fistula (with more than one cannulation)
* History of hematoma or stenosis in fistula
* Having an infection in the fistula area
* Taking painkillers 3 hours before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Invasive Pain at 12 Dialysis Session | At the end of the every dialysis session during one month (3 hemodialysis sessions are done every week)
  It will be assessed three times at the end of the dialysis session with Visual Analogue. Pain intensity measured on a Visual Analog Scale with scores ranging from 0 - 10. Pain increases as the score increases. The high point describes bad outcome.
Change From Baseline Post-Puncture Bleeding at 12 Dialysis Session | At the end of the every dialysis session during one month (3 hemodialysis sessions are done every week)
  Bleeding time was defined as the time (minutes) from the moment the pressure was applied to the moment when the bleeding stopped after the fistula needle was removed.

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crespo Montero R, Rivero Arellano F, Contreras Abad MD, Martinez Gomez A, Fuentes Galan MI. Pain degree and skin damage during arterio-venous fistula puncture. EDTNA ERCA J. 2004 Oct-Dec;30(4):208-12. doi: 10.1111/j.1755-6686.2004.tb00369.x. PMID 15835412
- [Background] Gaspar LJ, Moreira NM, Moutinho AA, Pinto PJ, Lima HB, Rodrigues F. Puncture of the arteriovenous fistula: bevel upward or bevel downward? EDTNA ERCA J. 2003 Apr-Jun;29(2):104. doi: 10.1111/j.1755-6686.2003.tb00284.x. No abstract available. PMID 14598956
- [Background] Marticorena RM, Donnelly SM. Impact of needles in vascular access for hemodialysis. J Vasc Access. 2016 Mar;17 Suppl 1:S32-7. doi: 10.5301/jva.5000534. Epub 2016 Mar 6. PMID 26951901